CLINICAL TRIAL: NCT06518265
Title: Osteosynthesis of High-Risk Ankle Fractures Using Locked Fibula Nails: What Results for Which Patients? A Monocentric Case Series
Brief Title: Osteosynthesis of High-Risk Ankle Fractures Using Locked Fibula Nails: What Results for Which Patients?
Acronym: OFCCF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A00925-42
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Ankle Fractures:Osteosynthesis of High-Risk Ankle Fractures Using Locked Fibula Nails

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ankle fractures are among the most common injuries in orthopedic and trauma surgery, accounting for 9% of all fractures. They can be classified into isolated malleolar fractures (internal and/or external), pilon fractures, and distal tibia fractures, which affect the entire distal part of the tibia, depending on whether they are intra-articular or extra-articular.

The aging of the population and the increase in survival of multiple trauma patients lead to an increase in ankle fractures with high skin risk, whether due to an open fracture, soft tissue injury (crush, dermabrasion, etc.). ) or a major risk of scarring (chronic venous insufficiency, lymphedema, unbalanced diabetes.

The fibula nail is a recent, minimally invasive osteosynthesis method whose results seem at least equivalent to those of screwed plate osteosynthesis in numerous series in the literature. The most commonly used and most studied fibula nail in the literature is the Acumed fibula nail. In recent literature, the use of the fibula nail in the fixation of tibial pilon fractures and/or fractures of the distal quarter of the leg is associated with satisfactory results.

The elements collected as part of this study could make it possible to validate the use of the fibula nail in the management strategy for these fractures and thus better codify and standardize practices in this restricted and complex area of traumatology.

DETAILED DESCRIPTION:
Ankle fractures represent one of the most common injuries in orthopedic and trauma surgery with an incidence of 9% of all fractures. We distinguish between isolated fractures of the malleolus (internal and/or external), fractures of the tibial pilon and the distal quarter of the leg which concern the entire distal part of the tibia depending on whether they are intra- or extra-articular. The aging of the population and the increase in survival of multiple trauma patients lead to an increase in ankle fractures with high skin risk, whether due to an open fracture, soft tissue injury (crush, dermabrasion, etc.). ) or a major risk of scarring (chronic venous insufficiency, lymphedema, unbalanced diabetes, etc.).

The classic management of fractures of the fibula (external malleolus) is based on open reduction-fixation using a screwed plate, made through a longitudinal incision. Restoring the length of the fibula contributes to the reduction of fractures of the tibial pilon. However, in patients at high skin risk, plate fixation increases tissue trauma and can lead to scar complications and infections.

The fibula nail is a recent, minimally invasive osteosynthesis method whose results seem at least equivalent to those of screwed plate osteosynthesis in numerous series in the literature [BÄCKER 2019]. The most commonly used and most studied fibula nail in the literature is the Acumed fibula nail. In recent literature, the use of the fibula nail in the fixation of tibial pilon fractures and/or fractures of the distal quarter of the leg is associated with satisfactory results.

If the fibula nail seems equivalent to the screwed plate in "classic" ankle fractures, we can wonder if its minimally invasive nature does not give it an advantage over the screwed plate in the fixation of ankle fractures. high skin risk. To our knowledge, few series have been published concerning this subpopulation at risk and for which the fibula nail represents an interesting alternative.

Likewise, although a biomechanical study showed a higher rate of torsional fracture after fibula nail fixation versus screwed plate, the results of fibula nail fixation in unstable ankle fractures appear equivalent to those of fixing by screwed plates. As the notion of stability of ankle fractures is not clearly defined in the literature, we will refer to tri-malleolar fractures, dislocated bi-malleolar fractures, tibial pilon fractures and fractures of the distal quarter of the leg as unstable fractures. As the notion of skin risk is not clearly defined in the literature, we will designate as skin risk patients presenting with acute traumatic tissue damage associated or not with an open fracture evaluated according to the Oestern and Tscherne classification as well as patients presenting with a skin disease. chronic such as lipodermatosclerosis, lymphedema, varicose or arterial ulcer and skin atrophy secondary to long-term corticosteroid therapy compromising the healing of a longitudinal incision next to the fibula.

Expected benefits:

The elements collected as part of this study could make it possible to validate the use of the fibula nail in the management strategy for these fractures and thus better codify and standardize practices in this restricted and complex area of traumatology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient at the time of injury
* Unstable fracture of one or both ankles: tri-malleolar fracture, distal quarter of the leg, tibial pilon.
* High skin risk (acute traumatic tissue injury associated or not with an open fracture evaluated according to the Oestern and Tscherne classification, chronic skin disease such as lipodermatosclerosis, lymphedema, varicose or arterial ulcer and skin atrophy secondary to corticosteroid therapy long course compromising the healing of a longitudinal incision next to the fibula).
* Standard preoperative x-ray image (ankle face and profile)
* Standard image post-operative x-rays (ankle face and profile)
* No opposition to participation in the study.

Exclusion Criteria:

* Pregnant, breastfeeding women.
* Subject under guardianship, curatorship, deprived of liberty or under the protection of justice.
* Subject who are cognitively incapable of answering the questionnaire.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This single-center observational study selects all patients treated in the orthopedics and traumatology department at Grenoble Alpes University Hospital between 01/01/2021 and 12/31/2023 for an unstable ankle fracture with high cutaneous risk.
  Epidemiological data, preoperative management, operative data and radiological criteria are collected and analyzed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical and radiological results of patients treated for fixation of an unstable ankle fracture with high cutaneous risk including a fibula nail without access to the fibular fracture site. | 1 year
  obtaining bone consolidation (healing) without cutaneous complications.

SECONDARY OUTCOMES:
Evaluation of the quality of the radiological reduction. | 1 year
  Radiological criteria of McLenann
Evaluation of clinical results | 1 year
  Clinical scores of EFAS
Evaluation of clinical results | 1 year
  Clinical scores of Olerud and Molander
Evaluation of clinical results | 1 year
  Clinical scores of Kitaoka hindfoot
Assessment of complications | 1 year
  Complications: re-intervention(s)
Assessment of complications | 1 year
  Complications: infection
Assessment of complications | 1 year
  Complications: healing disorders
Assessment of complications | 1 year
  Complications: secondary displacement
Assessment of complications | 1 year
  Complications: discomfort of osteosynthesis equipment

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble Alpes university Hospital,La tronche, La Tronche, France